CLINICAL TRIAL: NCT06341634
Title: Surveillance of Suicide Ideation in Adolescents (VISIA)
Acronym: VISIA
Status: Enrolling by invitation | Type: Observational
Sponsor: Servicio Gallego de Salud (Other Government)
Collaborators: University of Vigo (Other); Complejo Hospitalario Universitario de Vigo (Other); Complexo Hospitalario de Ourense (Other); Fundacin Biomedica Galicia Sur (Other)
Responsible Party: Principal Investigator, Alejandro Alberto García Caballero, Coordinator of Mental Health Prevention/Promotion Programs, Servicio Gallego de Salud
Other Study IDs: VISIA; TED2021-130747B-C22 (Other Grant/Funding Number: European Union); 3494130747-130747-28-521 (Other: Ministry of Science and Innovation)
Record Dates: First submitted 2023-11-20; First posted 2024-04-02 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Suicide; Distress, Emotional; Adolescent Behavior; Healthy
Keywords: Suicide Prevention; Distress, Emotional; Adolescent Behavior; Artificial Intelligence; Proteomics
MeSH Terms: conditions — Suicide; Adolescent Behavior; Suicide Prevention

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ideation: Patients with current suicidal ideation, recruited by staff doctors and psychologists from the child and adolescent psychiatry units of the Álvaro Cunqueiro Hospital in Vigo and the University Hospital Complex in Ourense, who have been deemed suitable for participation and have had the participation conditions explained to them and their parents, will undergo the following assessment protocol:
  Paykel scale Mini International Neuropsychiatric Interview (MINI) Strengths and Difficulties Questionnaire (SDQ) Mood and Feelings Questionnaire (MFQ) European Bullying Intervention Project Questionnaire (EBIP-Q) Problematic Internet Use Scale in Adolescents (EUPI-A) Millon Adolescent Clinical Inventory (MACI)
  Multimodal experimental battery:
  Recording of voice features Video recording of facial microexpression Registering of autobiographical texts Collecting of saliva samples
- Clinical Population: Psychological or psychiatric patients, devoid of suicidal ideation, recruited by staff doctors and psychologists from the child and adolescent psychiatry units of the Álvaro Cunqueiro Hospital in Vigo and the University Hospital Complex in Ourense, who have been deemed suitable for participation and have had the participation conditions explained to them and their parents, will undergo the following assessment protocol:
  Paykel scale Mini International Neuropsychiatric Interview (MINI) Strengths and Difficulties Questionnaire (SDQ) Mood and Feelings Questionnaire (MFQ) European Bullying Intervention Project Questionnaire (EBIP-Q) Problematic Internet Use Scale in Adolescents (EUPI-A) Millon Adolescent Clinical Inventory (MACI)
  Multimodal experimental battery:
  Recording of voice features Video recording of facial microexpression Registering of autobiographical texts Collecting of saliva samples
- General Population: Students with no known psychological or psychiatric issues, and free of suicidal ideation in the past year, recruited from schools among students who voluntarily agree to participate, and who have been deemed suitable for participation and have had the participation conditions explained to them and their parents, will undergo the following assessment protocol:
  Paykel scale Mini International Neuropsychiatric Interview (MINI) Strengths and Difficulties Questionnaire (SDQ) Mood and Feelings Questionnaire (MFQ) European Bullying Intervention Project Questionnaire (EBIP-Q) Problematic Internet Use Scale in Adolescents (EUPI-A) Millon Adolescent Clinical Inventory (MACI)
  Multimodal experimental battery:
  Recording of voice features Video recording of facial microexpression Registering of autobiographical texts Collecting of saliva samples

SUMMARY:
The goal of this observational study is to validate an AI algorithm's capability to differentiate the population with suicidal ideation from a control population using various multimodal variables, including voice analysis, facial emotions, natural language, and proteomics data.

The primary research question it aims to answer is:

Is it possible to identify suicidal ideation and suicide risk in adolescents early and non-intrusively using multimodal data analysis through digital instruments equipped with artificial intelligence?

Participants in this study will be asked to:

Complete psychometric instruments to establish a gold standard for detecting suicide risk and suicidal ideation.

Provide voice recordings, facial emotion data, and linguistic content in natural and specific contexts.

Participate in salivary proteomics data collection.

This study compares three distinct groups:

Ideation: Adolescent patients with current suicidal ideation. Clinical Population: Psychological or psychiatric patients of the same age and gender without suicidal ideation.

General Population: Adolescents without known psychological or psychiatric pathology of the same age and gender, without suicidal ideation.

Researchers will compare these groups to determine if the AI algorithm is effective in differentiating individuals with suicidal ideation (Group 1) from both a clinical control group (Group 2) and a general population control group (Group 3) using the collected multimodal data. The study aims to assess the algorithm's ability to identify early signs of suicide risk in these distinct participant populations.

DETAILED DESCRIPTION:
Introduction:

The Surveillance of Suicide Ideation in Adolescents (VISIA) project is a collaborative effort involving a diverse research team encompassing experts in mental disorders and seasoned researchers in data science, specializing in intelligent services and applications across various domains. The project aims to address the shortcomings identified in existing research. The initial phase of this endeavor seeks to validate an artificial intelligence (AI) algorithm capable of distinguishing individuals with suicidal ideation from a control group by analyzing multimodal variables. These variables include voice analysis, facial emotions, natural language, and proteomics. The cases will be labeled following established protocols.

Hypothesis:

The primary research question driving this project is: Can early and non-intrusive identification of suicidal ideation and suicide risk in young adults be achieved using multimodal data analysis through digital instruments equipped with artificial intelligence?

Objectives:

The overarching objective of this proposal is to design and implement an automated system for detecting emotional distress and suicide risk in adolescents aged between 11 and 16 using AI. This detection relies on molecular profiles derived from salivary proteomics, video and audio recordings in diverse contexts, and the linguistic content generated by the study participants. The integration of molecular profiles with data from video and audio recordings promises enhanced detection capabilities, providing a competitive edge in the development of future diagnostic tools.

Specific Objectives:

To realize the goals outlined above and tackle the scientific and technological challenges, the following specific objectives are established:

Development of a gold standard for detecting suicide risk and suicidal ideation in adolescents.

Identification of biomarkers (e.g., voice, facial expressions, salivary molecular fingerprint) relevant to characterizing adolescents with regard to suicide risk.

Identification of pertinent multimodal features for characterizing adolescents in relation to suicide risk.

Labeling of samples and AI model training.

Methodology:

Design and Study Subjects:

The study adopts a non-interventionist, analytical, observational, and prospective approach. It encompasses three distinct groups for comparison:

Ideation: Comprising individuals with current suicidal ideation. Clinical Population: Consisting of psychological or psychiatric patients of the same age and gender, devoid of suicidal ideation.

General Population: Encompassing adolescents with no known psychological or psychiatric issues, matched in age and gender, and free of suicidal ideation.

All three groups will undergo assessments using psychometric instruments, serving as a gold standard for AI system training and validation.

In summary, the VISIA project endeavors to leverage artificial intelligence and multimodal data analysis to detect suicidal ideation and suicide risk in adolescents, offering the potential for early and non-intrusive identification. The study's comprehensive methodology, involving diverse subject groups and rigorous data collection, is poised to contribute significantly to the field of mental health research and diagnostic tool development.

ELIGIBILITY:
Inclusion Criteria:

Ideation Group

* Participants must be between 11 and 16 years old.
* Patients who do not meet any of the exclusion criteria and whose parents (both), guardians, or legal representatives accept their voluntary participation in the study. In case of divorce, authorization from both parents will be required.
* Patients receive care in child and adolescent psychiatry or psychology services and currently have suicidal ideation.
* Patients may have a previous follow-up, as long as they have suicidal ideation at the present moment, or they may be new consultations and may be receiving pharmacological treatment (which will be documented in the study).

Clinical Population Group

* Participants must be between 11 and 16 years old.
* Patients who do not meet any of the exclusion criteria and whose parents (both), guardians, or legal representatives accept their voluntary participation in the study. In case of divorce, authorization from both parents will be required.
* Patients receive care in child and adolescent psychiatry or psychology services for any reason other than those listed as exclusion criteria.
* Patients have not had suicidal ideation in the past year. Patients may have a previous follow-up or may be new consultations, and they may be receiving pharmacological treatment (which will be documented in the study).

General Population Group

* Participants must be between 11 and 16 years old.
* Students who do not meet any of the exclusion criteria and whose parents (both), guardians, or legal representatives accept their voluntary participation in the study. In case of divorce, authorization from both parents will be required.
* Students must declare that they have not received psychiatric or psychological follow-up before, nor have they had suicidal ideation in the past year.

Exclusion Criteria (applicable to all groups):

* Neurodevelopmental disorders or speech disorders affecting verbal communication capacity, specifically including:
* Autism Spectrum Disorder grades 2 and 3.
* Communication disorders (selective mutism, language disorder, phonological disorder, childhood-onset fluency disorder, social communication disorder).
* Individuals with hearing impairment and verbal language impairment.
* Individuals with moderate and severe intellectual disabilities.
* Individuals with psychotic disorders.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescents aged between 11 and 16 years old from clinical and and general population.
Sampling Method: Non-Probability Sample
Enrollment: 339 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) | through study completion, an average of 1 year
  This questionnaire detects probable cases of mental and behavioral disorders in children and adolescents aged 4 to 17. A score >19 points is considered positive in screening.
Mood and Feelings Questionnaire (MFQ) | through study completion, an average of 1 year
  This questionnaire assesses symptoms of depression/suicide risk. Scores above 27 points are considered positive for screening. Higher values are indicative of worse outcomes.
Paykel Suicide Scale (PSS) | through study completion, an average of 1 year
  This questionnaire asks about suicidal ideation over the past year. Scores equal to or greater than 4 are suggestive of suicidal ideation. Higher values are indicative of worse outcomes.
Facial microexpressions, voice and linguistic content analysis | through study completion, an average of 1 year
  Participants will be asked to speak in front of a camera about their emotional state over the past week. The recording will have a minimum duration of 2 minutes and will be used for voice analysis, facial microexpressions, and natural language processing (NLP) for linguistic content analysis.
  Participants will also be asked to write a brief text on the computer in response to questions about how they perceive themselves and how they think others perceive them. The maximum duration for this exercise is 10 minutes.
Proteomic and stress level analysis | through study completion, an average of 1 year
  The collection of saliva is performed in a simple, non-invasive, and painless manner, allowing for the subsequent retrieval of high-quality proteins for further analysis and studies.

SECONDARY OUTCOMES:
Millon Adolescent Clinical Inventory - II (MACI-II) | through study completion, an average of 1 year
  A self-report questionnaire developed to evaluate the psychological functioning of adolescents. It assesses three domains in adolescent development. The average completion time is 30 minutes and can be conducted in groups.
Problematic Internet Use Scale in Adolescents (EUPI-A) | through study completion, an average of 1 year
  This 11-item questionnaire screens for problematic use of Internet among teenagers, ranginf fromm 0 to 44, with a cut-off for problematic use of 16 points. Higher values are indicative of worse outcomes.
European Bullying Intervention Project Questionnaire (EBIP-Q) and European Ciberbullying Intervention Project Questionnaire (ECIP-Q) | through study completion, an average of 1 year
  This tool for jointly assessing bullying and cyberbullying cointains The European Bullying Intervention Project Questionnaire (14-items) and the European Cyberbullying Intervention Project Questionnaire (22-items), both of Likert nature that respectively evaluate behaviors related to bullying and cyber-bullying. Higher values are indicative of worse outcomes.

OTHER OUTCOMES:
Oviedo Response Infrequency Scale-Revised (INF-OV-R) | through study completion, an average of 1 year
  Is a 10 items self-report measurement with a dichotomous response format (Yes/No) developed to detect those participants who respond randomly, pseudo-randomly, or dishonestly to the administered measuring instruments. The items on this scale are typically intermixed with questions and statements from other self-report measures that are administered together to o enable better detection. Higher values are indicative of random, pseudo-random, or dishonest answers.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro García Caballero, Principal Investigator — University Hospital Complex of Ourense
Locations (4):
- Spain (4):
  - Servizo Galego de Saúde, Santiago de Compostela, A Coruña
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - University of Vigo, Vigo, Pontevedra
  - University Hospital Complex of Ourense, Ourense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abd-Alrazaq AA, Alajlani M, Alalwan AA, Bewick BM, Gardner P, Househ M. An overview of the features of chatbots in mental health: A scoping review. Int J Med Inform. 2019 Dec;132:103978. doi: 10.1016/j.ijmedinf.2019.103978. Epub 2019 Sep 25. PMID 31622850
- [Background] Adamou M, Antoniou G, Greasidou E, Lagani V, Charonyktakis P, Tsamardinos I, Doyle M. Toward Automatic Risk Assessment to Support Suicide Prevention. Crisis. 2019 Jul;40(4):249-256. doi: 10.1027/0227-5910/a000561. Epub 2018 Nov 26. PMID 30474411
- [Background] Bachmann S. Epidemiology of Suicide and the Psychiatric Perspective. Int J Environ Res Public Health. 2018 Jul 6;15(7):1425. doi: 10.3390/ijerph15071425. PMID 29986446
- [Background] Briere J, Gil E. Self-mutilation in clinical and general population samples: prevalence, correlates, and functions. Am J Orthopsychiatry. 1998 Oct;68(4):609-20. doi: 10.1037/h0080369. PMID 9809120
- [Background] Brunner R, Kaess M, Parzer P, Fischer G, Carli V, Hoven CW, Wasserman C, Sarchiapone M, Resch F, Apter A, Balazs J, Barzilay S, Bobes J, Corcoran P, Cosmanm D, Haring C, Iosuec M, Kahn JP, Keeley H, Meszaros G, Nemes B, Podlogar T, Postuvan V, Saiz PA, Sisask M, Tubiana A, Varnik A, Wasserman D. Life-time prevalence and psychosocial correlates of adolescent direct self-injurious behavior: a comparative study of findings in 11 European countries. J Child Psychol Psychiatry. 2014 Apr;55(4):337-48. doi: 10.1111/jcpp.12166. Epub 2013 Nov 12. PMID 24215434
- [Background] Choi D, Sumner SA, Holland KM, Draper J, Murphy S, Bowen DA, Zwald M, Wang J, Law R, Taylor J, Konjeti C, De Choudhury M. Development of a Machine Learning Model Using Multiple, Heterogeneous Data Sources to Estimate Weekly US Suicide Fatalities. JAMA Netw Open. 2020 Dec 1;3(12):e2030932. doi: 10.1001/jamanetworkopen.2020.30932. PMID 33355678
- [Background] Krageloh CU, Czuba KJ, Billington DR, Kersten P, Siegert RJ. Using feedback from patient-reported outcome measures in mental health services: a scoping study and typology. Psychiatr Serv. 2015 Mar 1;66(3):224-41. doi: 10.1176/appi.ps.201400141. Epub 2014 Dec 1. PMID 25727110
- [Background] Gillies D, Christou MA, Dixon AC, Featherston OJ, Rapti I, Garcia-Anguita A, Villasis-Keever M, Reebye P, Christou E, Al Kabir N, Christou PA. Prevalence and Characteristics of Self-Harm in Adolescents: Meta-Analyses of Community-Based Studies 1990-2015. J Am Acad Child Adolesc Psychiatry. 2018 Oct;57(10):733-741. doi: 10.1016/j.jaac.2018.06.018. Epub 2018 Aug 21. PMID 30274648
- [Background] Coppersmith G, Leary R, Crutchley P, Fine A. Natural Language Processing of Social Media as Screening for Suicide Risk. Biomed Inform Insights. 2018 Aug 27;10:1178222618792860. doi: 10.1177/1178222618792860. eCollection 2018. PMID 30158822
- [Background] Czeisler ME, Lane RI, Petrosky E, Wiley JF, Christensen A, Njai R, Weaver MD, Robbins R, Facer-Childs ER, Barger LK, Czeisler CA, Howard ME, Rajaratnam SMW. Mental Health, Substance Use, and Suicidal Ideation During the COVID-19 Pandemic - United States, June 24-30, 2020. MMWR Morb Mortal Wkly Rep. 2020 Aug 14;69(32):1049-1057. doi: 10.15585/mmwr.mm6932a1. PMID 32790653
- [Background] Deveci A, Aydemir O, Taskin O, Taneli F, Esen-Danaci A. Serum BDNF levels in suicide attempters related to psychosocial stressors: a comparative study with depression. Neuropsychobiology. 2007;56(2-3):93-7. doi: 10.1159/000111539. Epub 2007 Nov 23. PMID 18037819
- [Background] Fernandez-Martinez I, Morales A, Mendez FX, Espada JP, Orgiles M. Spanish Adaptation and Psychometric Properties of the Parent Version of the Short Mood and Feelings Questionnaire (SMFQ-P) in a Non-Clinical Sample of Young School-Aged Children. Span J Psychol. 2020 Nov 5;23:e45. doi: 10.1017/SJP.2020.47. PMID 33148355
- [Background] Garcia de la Garza A, Blanco C, Olfson M, Wall MM. Identification of Suicide Attempt Risk Factors in a National US Survey Using Machine Learning. JAMA Psychiatry. 2021 Apr 1;78(4):398-406. doi: 10.1001/jamapsychiatry.2020.4165. PMID 33404590
- [Background] Golan O, Baron-Cohen S, Hill J. The Cambridge Mindreading (CAM) Face-Voice Battery: Testing complex emotion recognition in adults with and without Asperger syndrome. J Autism Dev Disord. 2006 Feb;36(2):169-83. doi: 10.1007/s10803-005-0057-y. PMID 16477515
- [Background] Hawgood J, De Leo D. Suicide Prediction - A Shift in Paradigm Is Needed. Crisis. 2016 Jul;37(4):251-255. doi: 10.1027/0227-5910/a000440. No abstract available. PMID 27809591
- [Background] Jacobson CM, Gould M. The epidemiology and phenomenology of non-suicidal self-injurious behavior among adolescents: a critical review of the literature. Arch Suicide Res. 2007;11(2):129-47. doi: 10.1080/13811110701247602. PMID 17453692
- [Background] Johnston JN, Campbell D, Caruncho HJ, Henter ID, Ballard ED, Zarate CA. Suicide Biomarkers to Predict Risk, Classify Diagnostic Subtypes, and Identify Novel Therapeutic Targets: 5 Years of Promising Research. Int J Neuropsychopharmacol. 2022 Mar 17;25(3):197-214. doi: 10.1093/ijnp/pyab083. PMID 34865007
- [Background] Kaess M, Parzer P, Haffner J, Steen R, Roos J, Klett M, Brunner R, Resch F. Explaining gender differences in non-fatal suicidal behaviour among adolescents: a population-based study. BMC Public Health. 2011 Jul 28;11:597. doi: 10.1186/1471-2458-11-597. PMID 21794184
- [Background] Kamali M, Saunders EF, Prossin AR, Brucksch CB, Harrington GJ, Langenecker SA, McInnis MG. Associations between suicide attempts and elevated bedtime salivary cortisol levels in bipolar disorder. J Affect Disord. 2012 Feb;136(3):350-8. doi: 10.1016/j.jad.2011.11.027. Epub 2011 Dec 10. PMID 22154566
- [Background] Karege F, Perret G, Bondolfi G, Schwald M, Bertschy G, Aubry JM. Decreased serum brain-derived neurotrophic factor levels in major depressed patients. Psychiatry Res. 2002 Mar 15;109(2):143-8. doi: 10.1016/s0165-1781(02)00005-7. PMID 11927139
- [Background] Kouter K, Videtic Paska A. 'Omics' of suicidal behaviour: A path to personalised psychiatry. World J Psychiatry. 2021 Oct 19;11(10):774-790. doi: 10.5498/wjp.v11.i10.774. eCollection 2021 Oct 19. PMID 34733641
- [Background] Lo Moro G, Soneson E, Jones PB, Galante J. Establishing a Theory-Based Multi-Level Approach for Primary Prevention of Mental Disorders in Young People. Int J Environ Res Public Health. 2020 Dec 16;17(24):9445. doi: 10.3390/ijerph17249445. PMID 33339317
- [Background] Meadows R, Hine C, Suddaby E. Conversational agents and the making of mental health recovery. Digit Health. 2020 Nov 20;6:2055207620966170. doi: 10.1177/2055207620966170. eCollection 2020 Jan-Dec. PMID 33282335
- [Background] Miranda-Mendizabal A, Castellvi P, Pares-Badell O, Alayo I, Almenara J, Alonso I, Blasco MJ, Cebria A, Gabilondo A, Gili M, Lagares C, Piqueras JA, Rodriguez-Jimenez T, Rodriguez-Marin J, Roca M, Soto-Sanz V, Vilagut G, Alonso J. Gender differences in suicidal behavior in adolescents and young adults: systematic review and meta-analysis of longitudinal studies. Int J Public Health. 2019 Mar;64(2):265-283. doi: 10.1007/s00038-018-1196-1. Epub 2019 Jan 12. PMID 30635683
- [Background] Navarro MC, Ouellet-Morin I, Geoffroy MC, Boivin M, Tremblay RE, Cote SM, Orri M. Machine Learning Assessment of Early Life Factors Predicting Suicide Attempt in Adolescence or Young Adulthood. JAMA Netw Open. 2021 Mar 1;4(3):e211450. doi: 10.1001/jamanetworkopen.2021.1450. PMID 33710292
- [Background] Nock MK, Kazdin AE. Examination of affective, cognitive, and behavioral factors and suicide-related outcomes in children and young adolescents. J Clin Child Adolesc Psychol. 2002 Mar;31(1):48-58. doi: 10.1207/S15374424JCCP3101_07. PMID 11845650
- [Background] Pacheco-Lorenzo MR, Valladares-Rodriguez SM, Anido-Rifon LE, Fernandez-Iglesias MJ. Smart conversational agents for the detection of neuropsychiatric disorders: A systematic review. J Biomed Inform. 2021 Jan;113:103632. doi: 10.1016/j.jbi.2020.103632. Epub 2020 Dec 2. PMID 33276112
- [Background] Pandey GN, Dwivedi Y, Rizavi HS, Ren X, Zhang H, Pavuluri MN. Brain-derived neurotrophic factor gene and protein expression in pediatric and adult depressed subjects. Prog Neuropsychopharmacol Biol Psychiatry. 2010 May 30;34(4):645-51. doi: 10.1016/j.pnpbp.2010.03.003. Epub 2010 Mar 20. PMID 20227453
- [Background] Pinon-Blanco A, Vergara-Moragues E, Fernandez-Martinez R, Gutierrez-Martinez O, Alvarez-Counago M, Martinez-Reglero C, Rivera-Baltanas T, Otero-Lamas F, Olivares-Diez J, Spuch-Calvar C. Effectiveness of the “Trisquel” board game intervention program for patients with schizophrenia spectrum disorders. Actas Esp Psiquiatr. 2020 Sep;48(5):209-219. Epub 2020 Sep 1. PMID 33210279
- [Background] Ramirez-Cifuentes D, Freire A, Baeza-Yates R, Punti J, Medina-Bravo P, Velazquez DA, Gonfaus JM, Gonzalez J. Detection of Suicidal Ideation on Social Media: Multimodal, Relational, and Behavioral Analysis. J Med Internet Res. 2020 Jul 7;22(7):e17758. doi: 10.2196/17758. PMID 32673256
- [Background] Rao ML, Hawellek B, Papassotiropoulos A, Deister A, Frahnert C. Upregulation of the platelet Serotonin2A receptor and low blood serotonin in suicidal psychiatric patients. Neuropsychobiology. 1998;38(2):84-9. doi: 10.1159/000026522. PMID 9732208
- [Background] Roe D, Mazor Y, Gelkopf M. Patient-reported outcome measurements (PROMs) and provider assessment in mental health: a systematic review of the context of implementation. Int J Qual Health Care. 2021 Mar 5;34(Suppl 1):ii28-ii39. doi: 10.1093/intqhc/mzz084. PMID 31725153
- [Background] Rothe J, Buse J, Uhlmann A, Bluschke A, Roessner V. Changes in emotions and worries during the Covid-19 pandemic: an online-survey with children and adults with and without mental health conditions. Child Adolesc Psychiatry Ment Health. 2021 Feb 21;15(1):11. doi: 10.1186/s13034-021-00363-9. PMID 33612122
- [Background] Spreux-Varoquaux O, Alvarez JC, Berlin I, Batista G, Despierre PG, Gilton A, Cremniter D. Differential abnormalities in plasma 5-HIAA and platelet serotonin concentrations in violent suicide attempters: relationships with impulsivity and depression. Life Sci. 2001 Jun 29;69(6):647-57. doi: 10.1016/s0024-3205(01)01158-4. PMID 11476186
- [Background] Tsui FR, Shi L, Ruiz V, Ryan ND, Biernesser C, Iyengar S, Walsh CG, Brent DA. Natural language processing and machine learning of electronic health records for prediction of first-time suicide attempts. JAMIA Open. 2021 Mar 17;4(1):ooab011. doi: 10.1093/jamiaopen/ooab011. eCollection 2021 Jan. PMID 33758800
- [Background] Vaidyam AN, Wisniewski H, Halamka JD, Kashavan MS, Torous JB. Chatbots and Conversational Agents in Mental Health: A Review of the Psychiatric Landscape. Can J Psychiatry. 2019 Jul;64(7):456-464. doi: 10.1177/0706743719828977. Epub 2019 Mar 21. PMID 30897957
- [Background] Vallejo-Curto MDC, Rodrigues-Amorim D, Jardon-Golmar L, Blanco-Formoso M, Rivera-Baltanas T, Rodriguez-Jamardo C, Fernandez-Palleiro P, Alvarez-Ariza M, Lopez-Garcia M, Garcia-Caballero A, de Las Heras E, Olivares JM, Spuch C. Proteomic and metabolic profiling of chronic patients with schizophrenia induced by a physical activity program: Pilot study. Rev Psiquiatr Salud Ment (Engl Ed). 2021 Jul-Sep;14(3):125-138. doi: 10.1016/j.rpsmen.2021.07.002. Epub 2021 Aug 10. PMID 34384726
- [Background] Voss C, Ollmann TM, Miche M, Venz J, Hoyer J, Pieper L, Hofler M, Beesdo-Baum K. Prevalence, Onset, and Course of Suicidal Behavior Among Adolescents and Young Adults in Germany. JAMA Netw Open. 2019 Oct 2;2(10):e1914386. doi: 10.1001/jamanetworkopen.2019.14386. PMID 31664450
- [Background] Zhang Y, Zhang O, Wu Y, Lee HJ, Xu J, Xu H, Roberts K. Psychiatric symptom recognition without labeled data using distributional representations of phrases and on-line knowledge. J Biomed Inform. 2017 Nov;75S:S129-S137. doi: 10.1016/j.jbi.2017.06.014. Epub 2017 Jun 15. PMID 28624644
- [Background] Rial Boubeta A, Gomez Salgado P, Isorna Folgar M, Araujo Gallego M, Varela Mallou J. PIUS-a: Problematic Internet Use Scale in adolescents. Development and psychometric validation. Adicciones. 2015 Mar 1;27(1):47-63. PMID 25879477
- [Background] Parkhi O., Vedaldi A., and Zisserman A.. 2015. Deep Face Recognition. In Proceedings of the British Machine Vision Conference (BMVC). 41.1-41.12.
- [Background] De Quiroga S, Riesgo M, Martín del Campo E, Pulido S, Rodrigo S. (2019) Impacto Socioeconómico de la depresión y el suicidio en España [Internet]. Rev Esp Econ Salud: 2019; 4(15).
- [Background] Stappen, L., Baird, A., Christ, L., Schumann, L., Sertolli, B., Messner, E., Cambria, E., Zhao, G., Schuller, Björn. (2021). The MuSe 2021 Multimodal Sentiment Analysis Challenge: Sentiment, Emotion, Physiological-Emotion, and Stress.
- [Background] Vekiri I. and Chronaki A. (2008) "Gender issues in technology use: Perceived social support, computer self-efficacy and value beliefs, and computer use beyond school," Comput. Educ., vol. 51, no. 3, pp. 1392-1404, 2008.
- [Background] World Health Organization (2014) Preventing suicide. A global imperative. Geneva: 2014.
- [Background] World Health Organisation (2021a) Comprehensive mental health action plan 2013-2030. Geneva: World Health Organization; 2021. Licence: CC BY-NC-SA 3.0 IGO.
- [Background] World Health Organisation (2021b) Suicide in the world: global health estimates. 2019, 32 p., World Health Organization, Technical documents. WHO/MSD/MER/19.3.
- See also: Suicide Risk Protocol — https://www.edu.xunta.gal/portal/sites/web/files/protocolo_risco_suicida-v.12.pdf